CLINICAL TRIAL: NCT01853826
Title: An Open Label Trial of Afatinib (Giotrif) in Treatment-naive (1st Line) or Chemotherapy Pre-treated Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring EGFR Mutation(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.55; 2009-017661-34 (EudraCT Number)
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- Afatinib treated-patients (Experimental): Patients diagnosed with EGFR mutation positive non-small cell lung cancer (NSCLC) locally advanced or metastatic who have never been treated with EGFR tyrosine kinase inhibitors (TKI) received a daily dose of 40 milligrams (mg) of afatinib (Giotrif®), in the form of film-coated tablet over a 28 day cycle. Afatinib was taken orally with 250 milliliters (mL) of water at the same time of the day and without eating anything for at least 3 hours. Patients continued on treatment for as long as there was no disease progression or no other trial withdrawal criteria. The dose was reduced to 30 mg or 20 mg once daily when the initial dose was not tolerated by the patient.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Patients received a daily dose of 40 milligrams (mg) of afatinib (Giotrif®), in the form of film-coated tablet over a 28 day cycle. Afatinib was taken orally with 250 milliliters (mL) of water at the same time of the day and without eating anything for at least 3 hours. Patients continued on treatment for as long as there was no disease progression or no other trial withdrawal criteria. The dose was reduced to 30 mg or 20 mg once daily when the initial dose was not tolerated by the patient.
  Other Names: Giotrif®

SUMMARY:
To evaluate the safety and tolerability of afatinib (Giotrif) in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR mutation(s) and have never been treated with an EGFR-TKI

ELIGIBILITY:
Inclusion criteria:

Patients with:

* locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC)
* Epidermal Growth Factor Receptor (EGFR) mutation-positive result per the institution's testing methodology.
* Adequate organ function, defined as all of the following:

  1. Absolute Neutrophil Count (ANC) > 1500/mm3. (ANC >1000/mm3 may be considered in special circumstances such as benign cyclical neutropenia as judged by the investigator and in discussion with the sponsor).
  2. Platelet count >75,000/mm3
  3. Serum creatinine < 1.5 times of the upper limit of normal
  4. Total Bilirubin < 1.5 times upper limit of (institutional) normal (Patients with Gilbert's syndrome total bilirubin must be <4 times institutional upper limit of normal).
  5. Aspartate Amino Transferase (AST) or Alanine Amino Transferase (ALT) < three times the upper limit of (institutional) normal (ULN) (if related to liver metastases < five times ULN).
* Eastern Cooperative Oncology Group (ECOG) score between 0 - 2
* written informed consent by patient or guardian prior to admission into the trial that is consistent with International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP) guidelines and local law.

Exclusion criteria:

Patients who or with:

* prior treatment with an EGFR tyrosine kinase inhibitor (TKI)
* anti-cancer treatment within 2 weeks prior to start of trial treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted)
* radiotherapy within 14 days prior to drug administration, except as follows:

  1. Palliative radiation to organs other than chest may be allowed up to 2 weeks prior to drug administration, and
  2. Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
* previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* known pre-existing interstitial lung disease
* meningeal carcinomatosis and symptomatic brain metastases (patients with asymptomatic brain metastases, who were previously treated, are eligible provided they have had Stable Disease (SD) for at least 4 weeks on stable doses of medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (118):
- Australia (3):
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Sunshine Hospital, AT Albans, Victoria
  - St John of God Murdoch, Murdoch, Western Australia
- Austria (4):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - Klinik Penzing SMZ Baumgartner Hoehe, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- Czechia (4):
  - University Hospital Brno, Brno
  - Hospital Hradec Kralove, Hradec Králové
  - University Hospital Ostrava, Ostrava
  - University Hospital Plzen, Plzen-Bory, Pilsen
- Greece (4):
  - Chest Hospital of Athens "Sotiria", Athens
  - Metropolitan Hospital, Oncology Clinic, N. Faliro
  - General Oncology Hospital "Agioi Anargyri", Nea Kifissia
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Hungary (4):
  - Koranyi National Institute For Pulmonolgy, Budapest
  - Institute of Chest Diseases Csongrad County,Dpt. Pulmonology, Deszk
  - Pulmonology Institute of Veszprem County, Farkasgyepu, Farkasgyepü
  - Fejer County Saint George University Teaching Hospital, Székesfehérvár
- Israel (5):
  - Soroka Univ. Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center Tel HaShomer, Tel Litwinsky
- Italy (44):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Az. Ospedaliere Umberto I di Ancona, Ancona
  - A. O. Giuseppe Moscati, Avellino
  - Centro di riferimento Oncologico, Aviano (PN)
  - Istituto Tumori Giovanni Paolo II, Bari
  - A. O. Ospedali Riuniti di Bergamo, Bergamo
  - Policlinico S. Orsola Malpighi, Bologna
  - Ospedale Centrale di Bolzano, Bolzano
  - A.O. Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Careggi, Florence
  - Azienda Ospedaliera San Martino, Genova
  - Osp. S. Maria della Scaletta, Imola
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Osp. Campo di Marte, Lucca
  - Istituto Scientifico Romagnolo, Meldola (FC)
  - IRCCS Fondazione Ospedale Maggiore, Milan
  - IRCCS San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Università di Modena e Reggio Emilia, Modena
  - A.O. San Gerardo di Monza, Monza (MI)
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - Osp. dei Colli Monaldi-Cotugno, Napoli
  - A.O.U. Maggiore della Carita', Novara
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano (TO)
  - Istituto Oncologico Veneto IRCCS, Padua
  - A.O. Univ. Policlinico "Paolo Giaccone", Palermo
  - Casa di Cura La Maddalena, Palermo
  - Azienda Ospedaliera di Parma, Parma
  - Ospedale S.Maria della Misericordia, AO di Perugia, Perugia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Ospedale S. Maria delle Croci, Ravenna
  - Irccs Crob, Rionero in Vulture (PZ)
  - Università Campus Bio-Medico - ROMA, Roma
  - Istittuo Nazionale Tumori Regina Elena - IRCCS, Roma
  - A.O. San Camillo Forlanini, Roma
  - Poli Univ A. Gemelli, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera "Santo Maria", Terni
  - AO Città della Salute e Scienza, Torino
  - Ospedale S. Maria di Ca' Foncello Azienda ULSS9 TREVISO, Treviso
  - A. O. S. Maria della Misericordia, Udine
  - Ospedale Policlinico G.B. Rossi (Borgo Roma) di Verona, Verona
- Poland (6):
  - Oncology Center na F. Lukaszczyka, Bydgoszcz
  - University Clinical Center, Gdansk, Gdansk
  - Provincial Specialist M. Kopernik Hospital, Lodz
  - MS Clinsearch, Private Practice, Lublin
  - MED POLONIA SP Z O O, Clinical Trials Department,Poznan, Poznan
  - Oncology Center-Maria Sklodowska-Curie Institute, Warsaw
- Portugal (5):
  - ULS de Coimbra, E.P.E., Coimbra
  - IPO Lisboa Francisco Gentil, EPE, Lisbon
  - Centro Hospitalar Lisboa Norte Hospital Pulido Valente, Lisbon
  - IPO Porto Francisco Gentil, EPE, Porto
  - ULS de Gaia/Espinho, EPE, Vila Nova de Gaia
- Russia (6):
  - St.Auton.Heal.Inst."Rep.Clin.Onc.Disp.of MoH of Rep. Tatarstan", Kazan'
  - Moscow City Oncology Dispensary, Moscow, Moscow
  - FSBI "N.N Blokhin Med.Res.Cent.Onc."MoH of RF, Moscow
  - Clinical Oncology Center, Omsk
  - St. Petersburg GUZ City Clinical Oncology Dispensary, Saint Petersburg
  - FSBI "N.N. Petrov National Medical Research Center of Oncology" of MoH of RF, Saint Petersburg
- Spain (33):
  - Hospital A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario de Cruces, Barakaldo (Bilbao)
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital de Canarias, La Laguna - Tenerife
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Puerta de Hierro, Majadahonda (Madrid)
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Politècnic La Fe, Valencia
  - Hospital Clínico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, multicentre, single-arm trial to evaluate the safety, tolerability and efficacy of afatinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) mutation(s) who had never been treated with an EGFR tyrosine kinase inhibitor (TKI).
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Afatinib Treated-patients
Started | 481
Treated | 479
Completed | 0
Not Completed | 481
Not completed — Patients who switched to commercial drug | 11
Not completed — Patient refused to continue medication | 21
Not completed — Lost to Follow-up | 2
Not completed — Non-compliant with protocol | 4
Not completed — Other adverse events (AE) | 62
Not completed — Worsening or AE of underlying cancer disease | 24
Not completed — Progressive disease | 342
Not completed — Other than listed | 13
Not completed — Not treated - not signed privacy informed consent | 2

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients who were dispensed afatinib and are documented to have taken at least one dose of afatinib.
Arm/Group | Afatinib Treated-patients
Number analyzed (Participants) | 479
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314
  Male | 165
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 465
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events According to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Number of patients with any treatment emergent adverse event (AE) according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: From first drug administration to last drug administration plus 28 days of residual effect period. Up to 3866 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib Treated-patients
Number analyzed (Participants) | 479
Participants | 478

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events and other AEs: From first drug administration to last drug administration plus 28 days of residual effect period. Up to 3866 days.
Description: Treated set (TS): all patients who were dispensed afatinib and are documented to have taken at least one dose of afatinib.
Arm/Group | Afatinib Treated-patients
All-Cause Mortality (participants affected / at risk) | 127/479
Serious Adverse Events (participants affected / at risk) | 210/479
Other Adverse Events (participants affected / at risk) | 268/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Treated-patients (N=479)
Coagulopathy (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Left ventricular dilatation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ventricular hypokinesia (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 16
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Gastric perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Intestinal infarction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Odynophagia (Gastrointestinal disorders) | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 3
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 2
Death (General disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 11
Hyperpyrexia (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Abscess (Infections and infestations) | 1
Abscess neck (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cavernous sinus thrombosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Clostridial infection (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Ear infection bacterial (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Viral infection (Infections and infestations) | 1
Accidental poisoning (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 2
Craniofacial fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 3
Hip fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian granulosa cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 5
Cerebrovascular disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 4
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 3
Ischaemic stroke (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Device dislocation (Product Issues) | 1
Behaviour disorder (Psychiatric disorders) | 1
Bradyphrenia (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 8
Urinary retention (Renal and urinary disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Surgery (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 4
Haematoma (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Treated-patients (N=479)
Diarrhoea (Gastrointestinal disorders) | 238
Nausea (Gastrointestinal disorders) | 32
Stomatitis (Gastrointestinal disorders) | 42
Asthenia (General disorders) | 52
Fatigue (General disorders) | 35
Mucosal inflammation (General disorders) | 54
Pyrexia (General disorders) | 30
Conjunctivitis (Infections and infestations) | 41
Paronychia (Infections and infestations) | 85
Decreased appetite (Metabolism and nutrition disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 28
Dry skin (Skin and subcutaneous tissue disorders) | 49
Pruritus (Skin and subcutaneous tissue disorders) | 29
Rash (Skin and subcutaneous tissue disorders) | 143
Rash papular (Skin and subcutaneous tissue disorders) | 27
Skin fissures (Skin and subcutaneous tissue disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT01853826/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT01853826/SAP_001.pdf